CLINICAL TRIAL: NCT07112573
Title: Association Between Intake of Psychotropic Medications and Risk of Falls in Older Adults
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD 139/2025
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-07

CONDITIONS: Falls (Accidents) in Old Age; Psychotropic Drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the association between intake of psychotropic medications and increased risk of falls in older adults discharged from Ain Shams University Geriatric Hospital as a primary outcome and incident fractures that may occur as a secondary outcome of such fall.

DETAILED DESCRIPTION:
The aim of the study is to assess the association between intake of psychotropic medications and increased risk of falls in older adults discharged from Ain Shams University Geriatric Hospital as a primary outcome and incident fractures that may occur as a secondary outcome of such fall. A prospective cohort study will be conducted. Older adults both males and females who were admitted to Ain Shams University, Geriatric Hospital will be included in this study with exclusion to patients with malignancy and bedridden patients. Baseline data will be collected retrospectively from the medical records of the patients admitted to Ain Shams University Geriatric Hospital from July 2024 till June 2025. Data include socio-demographic data, drug history, compliance on medications which will be assessed by Hill-Bone Medication Adherence Scale, history of falls, cognitive, psychological, nutritional and functional assessment and labs. Then follow up participants after 1 year after discharge from hospital through telephone call for occurrence of falls.

ELIGIBILITY:
Inclusion Criteria:

* patients (males and females) aged ≥ 60 years old patients who accept to participate in the study

Exclusion Criteria:

* Patients with malignancy Bedridden patients

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: older adults both males and females who were admitted to Ain Shams University, Geriatric Hospital
Sampling Method: Probability Sample
Enrollment: 398 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Association between intake of psychotropic medications and increased risk of falls in older adults | 1 year after discharge from hospital
  1. Association between positive history of intake of any psychotropic medication in the previous year and history of falls in the same year.
  2. Association between incidence of falls and duration of intake of psychotropic medications.
  3. Association between incidence of falls and the class of psychotropic medication(s) used.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt